CLINICAL TRIAL: NCT04310345
Title: Exploring the Impact of Human-Animal Interactions on Children With Life-Threatening Conditions and Their Parents
Brief Title: Impact of Human-Animal Interactions on Children With Life-Threatening Conditions and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maryjo Gilmer, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC PED 2003; R21HD097757-01 (NIH)
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Advanced Cancer; Relapsed Cancer; Refractory Cancer
MeSH Terms: conditions — Recurrence; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Animal-Assisted Interaction (Experimental): Children and their caregivers will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
  Interventions: Behavioral: Animal-Assisted Interactions

INTERVENTIONS:
Behavioral: Animal-Assisted Interactions — Child and caregivers will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.

SUMMARY:
This study will evaluate the effects of human-animal interaction on reducing anxiety, depression, worry, and pain and enhancing quality of life in children ages 6-17 years old with a life threatening cancer and their parent caregivers.

DETAILED DESCRIPTION:
Objectives:

* To examine the feasibility of human-animal interaction (HAI) sessions for children with a life threatening cancer and a primary caregiver, specifically to:

  * To identify and document necessary modifications for a safe and feasible intervention
  * To obtain recruitment estimates and determine potential recruitment barriers
  * To evaluate elements of implementation fidelity (design, training, delivery/receipt of treatment, enactment)
  * To verify safety
* To determine the preliminary efficacy of human-animal interaction sessions:

  * On children with a life threatening cancer for the outcomes of qualify of life, anxiety, depression, worry, and pain
  * On caregivers of children with a life threatening cancer for the outcomes of stress and anxiety

Exploratory Objective:

- To explore mechanisms (reduced salivary cortisol and urinary norepinephrine levels) associated with 8 weeks of human-animal interaction.

ELIGIBILITY:
Inclusion Criteria:

Child:

* Children age 6-17 years old that have been diagnosed with advanced cancer as defined by any stage of relapsed, recurrent or refractory cancer
* Able to understand English or Spanish to complete consents and surveys

Parent or Guardian:

* Parent or guardian as determined by person who brings child to >50% of their clinic visits
* Able to understand English or Spanish to complete consents and surveys

Exclusion Criteria for both Children and Parent/Guardian:

* Self-reported fear of or allergies to canines
* Cognitive impairment as identified by healthcare team or inability to complete consenting process

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryjo Gilmer, PhD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Animal-Assisted Interaction -- Child Participants: Children will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
  Animal-Assisted Interactions: Child will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
- Animal-Assisted Interaction -- Adult Participants: Caregivers will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
  Animal-Assisted Interactions: Caregivers will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
Period: Overall Study
Arm/Group | Animal-Assisted Interaction -- Child Participants | Animal-Assisted Interaction -- Adult Participants
Started | 31 | 43
Completed | 28 | 39
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Population: Children ages 6-17 years with advanced cancer and their parents were enrolled in the study. Measures of stress, anxiety, and quality of life were collected at baseline.
Groups:
- Animal-Assisted Interaction - Child Participants: Children will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
  Animal-Assisted Interactions: Child will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
- Animal-Assisted Interaction - Caregiver Participants: Caregivers will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
  Animal-Assisted Interactions: Caregivers will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital.
- Total: Total of all reporting groups
Arm/Group | Animal-Assisted Interaction - Child Participants | Animal-Assisted Interaction - Caregiver Participants | Total
Number analyzed (Participants) | 31 | 43 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 0 | 31
  Between 18 and 65 years | 0 | 43 | 43
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 28 | 41
  Male | 18 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 1 | 1 | 2
  White | 25 | 30 | 55
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 9 | 10
Region of Enrollment [Number; unit: participants]
  United States | 31 | 43 | 74

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Quality of Life
Description: The Pediatric Quality of Life Inventory (PedsQL) was administered to children and their parents (proxy for child quality of life) at baseline, week 4, and week 8 visits. Weeks 4 and 8 were after interacting with a therapy dog. Baseline surveys collected without seeing a therapy dog. The PedsQL Measurement is a validated scale to assess health-related quality of life in children and adolescents with acute and chronic health conditions. Scores are scaled from 1-100, with higher scores indicative of better quality of life.
Time Frame: Up to 2 months
Population: Children ages 6-17 with relapsed or refractory cancer and their caregivers who participated in therapy dog visits for up to 8 weeks at clinic visits or in the hospital.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Animal-Assisted Interaction - Child Participants (Baseline): Child will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital for up to 8 weeks. Baseline visit data on quality of life obtained through PedsQL survey without seeing therapy dog.
- Animal-Assisted Interaction - Child Participants (Week 4): Child will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital for up to 8 weeks. Week 4 data PedsQL survey conducted after seeing therapy dog.
- Animal-Assisted Interaction - Child Participants (Week 8): Child will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital for up to 8 weeks. Week 8 data PedsQL survey conducted after seeing therapy dog.
- Animal-Assisted Interaction - Caregiver Participants (Baseline): Caregivers will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital. Caregiver-Proxy data on child quality of life obtained using PedsQL survey. Baseline data obtained without seeing therapy dog.
- Animal-Assisted Interaction - Caregiver Participants (Week 4): Caregivers will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital. Caregiver-Proxy data on child quality of life obtained using PedsQL survey. Week 4 data obtained after seeing therapy dog.
- Animal-Assisted Interaction - Caregiver Participants (Week 8): Caregivers will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital. Caregiver-Proxy data on child quality of life obtained using PedsQL survey. Week 8 data obtained after seeing therapy dog.
Arm/Group | Animal-Assisted Interaction - Child Participants (Baseline) | Animal-Assisted Interaction - Child Participants (Week 4) | Animal-Assisted Interaction - Child Participants (Week 8) | Animal-Assisted Interaction - Caregiver Participants (Baseline) | Animal-Assisted Interaction - Caregiver Participants (Week 4) | Animal-Assisted Interaction - Caregiver Participants (Week 8)
Number analyzed (Participants) | 29 | 29 | 29 | 21 | 21 | 21
score on a scale
  PedsQL (Physical) | 47.6 (18.1) | 50.3 (23.5) | 61.6 (27.7) | 41.5 (24.1) | 37.8 (18.8) | 47.8 (24.7)
  PedsQL (Emotional) | 65.6 (20.6) | 65.7 (19.0) | 71.3 (20.1) | 51.9 (16.1) | 53.8 (18.4) | 58.8 (15.1)
  PedsQL (Social) | 72.5 (21.6) | 66.7 (23.1) | 66.7 (25.1) | 63.8 (20.5) | 61.4 (17.8) | 62.9 (20.7)
  PedsQL (School) | 48.0 (22.4) | 50.0 (21.3) | 56.7 (25.4) | 46.4 (19.2) | 50.5 (23.4) | 58.8 (21.8)
  PedsQL (Psycho-Social) | 64.1 (17.5) | 64.9 (18.6) | 69.6 (20.0) | 52.3 (16.0) | 54.4 (17.0) | 60.5 (13.9)
  PedsQL (Overall) | 55.7 (14.7) | 56.9 (18.2) | 64.7 (19.5) | 47.1 (15.9) | 47.5 (16.0) | 55.0 (15.1)

2. Primary Outcome: Anxiety
Description: The state-trait anxiety inventory State sub scale was administered to children (STAI-Child) and their parents (STAI) at baseline, week 4, and week 8. The 20-item STAI-CH is a validated scale for anxiety in children aged 5-17; the 20-item STAI is validated to assess anxiety in adult participants. The State subscale is intended to assess level of anxiety at the time of survey administration. Possible range of scores of the STAI-CH State subscale is 20-60, while the possible range from the STAI state subscale for adults is 20-80. Higher scores are indicative of increased anxiety. Baseline data were obtained without seeing a therapy dog, whereas STAI-CH and STAI surveys were conducted after seeing the therapy dog at weeks 4 and 8.
Time Frame: Up to 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Animal-Assisted Interaction - Child Participants (Baseline): Child will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital for up to 8 weeks. Baseline visit data on anxiety obtained through STAI-CH survey without seeing therapy dog.
- Animal-Assisted Interaction - Child Participants (Week 4): Child will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital for up to 8 weeks. Week 4 data STAI-CH survey conducted after seeing therapy dog.
- Animal-Assisted Interaction - Child Participants (Week 8): Child will spend approximately 10-15 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital for up to 8 weeks. Week 8 data STAI-CH survey conducted after seeing therapy dog.
- Animal-Assisted Interaction - Caregiver Participants (Baseline): Caregivers will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital. Caregiver data on anxiety obtained using STAI survey. Baseline data obtained without seeing therapy dog.
- Animal-Assisted Interaction - Caregiver Participants (Week 4): Caregivers will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital. Caregiver data on anxiety obtained using STAI survey. Week 4 data obtained after seeing therapy dog.
- Animal-Assisted Interaction - Caregiver Participants (Week 8): Caregivers will spend approximately 10-5 minutes with a registered canine and its owner during potentially anxiety-producing visits to the clinic or hospital. Caregiver data on anxiety obtained using STAI survey. Week 8 data obtained after seeing therapy dog.
Arm/Group | Animal-Assisted Interaction - Child Participants (Baseline) | Animal-Assisted Interaction - Child Participants (Week 4) | Animal-Assisted Interaction - Child Participants (Week 8) | Animal-Assisted Interaction - Caregiver Participants (Baseline) | Animal-Assisted Interaction - Caregiver Participants (Week 4) | Animal-Assisted Interaction - Caregiver Participants (Week 8)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29 | 29
units on a scale | 31.4 (5.2) | 29.2 (4.5) | 29.5 (5.8) | 40.2 (11.9) | 35.6 (10.9) | 35.9 (11.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the time frame each participant was assessed in relation to baseline which was a duration of up to 8 weeks.
Arm/Group | Animal-Assisted Interaction
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04310345/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04310345/ICF_000.pdf